CLINICAL TRIAL: NCT00505466
Title: Transition From Research to Disclosure in Human Genetics
Status: Completed | Type: Observational
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: BS99-038
Record Dates: First submitted 2007-07-19; First posted 2007-07-23 (Estimated); Last update posted 2022-03-04 (Actual); Status verified 2022-03

CONDITIONS: Education
Keywords: Human Genetics; Genetic Counseling; Genetic Testing; p53 Mutation; Genetics
MeSH Terms: interventions — Genetic Counseling

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Optional small sample of blood (about 6 tablespoons) for genetic testing for p53 following pre-test genetic counseling.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pre-Test Genetic Counseling + Genetic Sample
  Interventions: Behavioral: Genetic Counseling

INTERVENTIONS:
Behavioral: Genetic Counseling — Genetic counseling conducted in person, by telephone with an M. D. Anderson Genetic Counselor, or with a local Genetic Counselor in conference with the M. D. Anderson Genetic Counselor.

SUMMARY:
The goal of this study is to design a means of providing research families, from diverse geographical locations, the chance to receive genetic testing after having been educated by video, and meetings or telephone conversations with a genetic counselor/study professional.

This is an investigational study. About 800 people will be offered genetic testing. This study is being performed only at MD Anderson.

DETAILED DESCRIPTION:
Participants will receive pre-test genetic counseling in one of three ways: (1) in person at MD Anderson; (2) by telephone with an MD Anderson Genetic Counselor/study professional; (3) with a local Genetic Counselor in conference with the MD Anderson Genetic Counselor/study professional. After receiving pre-test genetic counseling, participants will be given the opportunity to schedule a submission of a small sample of blood (about 6 tablespoons) for genetic testing for p53. You may have this blood test repeated if there are any problems in the lab. The study doctor will discuss this with you.

Participants who submit a sample may choose to see a genetic counselor/study professional in person or schedule a phone conversation to receive the results of the genetic test. Genetic counseling may take place at MD Anderson at no cost. Participants may wish to have counseling close to their home, though they then are responsible for the cost of the counseling. If, after talking to the counselor/study professional, the participant wants to know the results of the test, he or she will be told. A participant will be given more counseling and advice on what other care might be needed and what other actions they should take.

The test results will be kept private. Names will not be used in computer records.

ELIGIBILITY:
Inclusion Criteria:

2.0 Genetic testing

Members of families who have participated in the p53 project through Dr. Strong's lab are eligible, via protocol P90-001. There are at least 145 kindreds including at least 800 participants living who may be at risk of carrying a p53 germline mutation. The participants must provide an informed consent and be 18 years or older. We will include English and non-English speaking participants. For non-English speaking participants to be recruited, the consent documents has been translated into the language of the target population in accordance with the IRB procedures.

2.1 Parents Attitudes toward testing children at risk for TP53 mutations

For the survey portion of this study, we will invite individuals who 1) are already enrolled in the P90-001 study), 2) have been known to carry a germline p53 mutation, and 3) have children who are less than 27 years old. Patients who agree to enroll in the survey portion of the study will be presented with a consent statement and a printed copy of the survey along with a postage-paid envelope which they can return (either by mail or in person) at their convenience.

2.2 Psychosocial impact of participating in LFS screening

1. Adults who have undergone genetic testing and have a confirmed p53 mutation
2. Adults participating in LFS screening program

Exclusion Criteria:

N/A

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patient diagnosed with cancer or a participant with a family member who has had cancer.
Sampling Method: Non-Probability Sample
Enrollment: 577 (Actual)
Dates: Start 1999-05-06 (Actual); Primary Completion 2022-02-08 (Actual); Study Completion 2022-02-08 (Actual)

PRIMARY OUTCOMES:
Number of Participants Received Pre-test Genetic Counseling | 10 Years

SECONDARY OUTCOMES:
Number of participants completing genetic testing for p53 | Baseline to time of follow-up (2 weeks, 6, and 12 months)

CONTACTS AND LOCATIONS:
Overall Officials: Louise C. Strong, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org